CLINICAL TRIAL: NCT06857331
Title: Optimization of Perioperative Analgesia With Erector Spinae Plane Block During Major Abdominal Surgeries in Patients With Impaired Liver Function
Brief Title: Perioperative Analgesia With Erector Spinae Plane Block in Liver Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Nazarii Mysynchuk, MD, Bogomolets National Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Liver Transplant; Erector Spina Plan Block
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liver transplant recipients without regional anesthesia (No Intervention): Liver transplant recipients without regional anesthesia
- Liver transplant recipients with regional anesthesia (ESP) (Experimental): ESP bilateral thoracic with a subsequent catheterization.
  Interventions: Procedure: Erector Spinae Plane Block using 0.2% ropivacaine

INTERVENTIONS:
Procedure: Erector Spinae Plane Block using 0.2% ropivacaine — Bilateral thoracic ESP block on the day of the transplantation with a subsequent catheterization will be suggested for the patients. In case of their written consent for the participation in the study this procedure will be performed on the day of the operation. 0.2% ropivacaine is going to be used throughout all the perioperative period.
  Arms: Liver transplant recipients with regional anesthesia (ESP)

SUMMARY:
The goal of this clinical trial is to learn if ESP block is safe and effective for perioperative analgesia in patients undergoing liver transplant. The main question it aims to answer are Is ESP block safe and has a minimum side effects, like hematoma? Is it effective for perioperative analgesia? Researchers will compare the results to a group of patients who underwent liver transplants without any regional anaesthesia techniques.

Participants will receive bilateral thoracic ESP block on the day of the transplantation with a subsequent bilateral catheterization.

ELIGIBILITY:
Inclusion Criteria:

* impaired liver function - cirrhosis or chronic liver disease with the development of hypocoagulation (APTT > 35 sec, INR > 1.5), thrombocytopenia, patients requiring major abdominal surgery, age > 18 years, written consent to participate in the study was obtained

Exclusion Criteria:

* Platelet count <50x109, failed ESP catheterization unilateral or bilateral, failed epidural anesthesia attempt, history of allergy or hypersensitivity to local anesthetics, hepatopulmonary syndrome, patients on mechanical ventilation before surgery, patients on CRRT before surgery, refusal to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Pain reduction postoperative | from enrollment to the 2nd postoperative day
  Pain assessment with scores
Opioid reduction intraoperatively | from enrollment to the end of the operation
  The amount of intraoperative fentanyl
Need for opioids postoperatively | from enrollment to the 2nd postoperative day
  Need for opioids postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Universal Hospital Oberig, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No